CLINICAL TRIAL: NCT04924062
Title: A Phase 3 Randomized, Double Blind Study of Pembrolizumab Plus Gemcitabine/Cisplatin Versus Placebo Plus Gemcitabine/Cisplatin as First-Line Therapy in Participants With Advanced and/or Unresectable Biliary Tract Carcinoma
Brief Title: Pembrolizumab (MK-3475) Plus Gemcitabine/Cisplatin Versus Placebo Plus Gemcitabine/Cisplatin for First-Line Advanced and/or Unresectable Biliary Tract Carcinoma (BTC) (MK-3475-966/KEYNOTE-966)-China Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3475-966 China Extension; MK-3475-966 (Other: MSD); KEYNOTE-966 (Other: MSD); 195007 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2021-06-08; First posted 2021-06-11 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Biliary Tract Carcinoma
Keywords: Programmed cell death 1 (PD-1); Pembrolizumab; Cholangiocarcinoma; Gallbladder cancer; Checkpoint inhibitor; Immunotherapy; Biliary; Keytruda; Bile Duct Cancer
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body; Cholangiocarcinoma; Gallbladder Neoplasms; Bile Duct Neoplasms | interventions — pembrolizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (Pembrolizumab+Gemcitabine+Cisplatin) (Experimental): Pembrolizumab, 200 mg, every 3 weeks (Q3W), Day 1 of each 3-week cycle for up to 35 cycles PLUS Gemcitabine, 1000 mg/m^2, Q3W, Day 1 and Day 8 of each cycle until progressive disease or unacceptable toxicity PLUS Cisplatin, 25 mg/m^2, Q3W, Day 1 and Day 8 of each cycle for up to 8 cycles.
  Interventions: Biological: Pembrolizumab; Drug: Gemcitabine; Drug: Cisplatin
- Arm B (Placebo+Gemcitabine+Cisplatin) (Placebo Comparator): Placebo to Pembrolizumab, 200 mg, every 3 weeks (Q3W), Day 1 of each 3-week cycle for up to 35 cycles PLUS Gemcitabine, 1000 mg/m^2, Q3W, Day 1 and Day 8 of each cycle until progressive disease or unacceptable toxicity PLUS Cisplatin, 25 mg/m^2, Q3W, Day 1 and Day 8 of each cycle for up to 8 cycles.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Placebo

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab by intravenous (IV) infusion
  Other Names: MK-3475
  Arms: Arm A (Pembrolizumab+Gemcitabine+Cisplatin)
Drug: Gemcitabine — Gemcitabine by IV infusion
  Other Names: Gemzar
Drug: Cisplatin — Cisplatin by IV infusion
  Other Names: Platinol®; Platinol®-AQ
Drug: Placebo — Placebo to pembrolizumab
  Arms: Arm B (Placebo+Gemcitabine+Cisplatin)

SUMMARY:
In this China Extension study, pembrolizumab plus gemcitabine/cisplatin will be compared with placebo plus gemcitabine/cisplatin as first-line therapy in Chinese adults with advanced and/or unresectable biliary tract carcinoma. The primary hypothesis is pembrolizumab plus gemcitabine/cisplatin is superior to placebo plus gemcitabine/cisplatin with respect to overall survival (OS).

DETAILED DESCRIPTION:
The China extension study will include participants previously enrolled in China in the global study for MK-3475-966 (NCT04003636) plus those enrolled during the China extension enrollment period. A total of approximately 158 Chinese participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria

* Has histologically confirmed diagnosis of advanced (metastatic) and/or unresectable (locally advanced) biliary tract cancer (intra-or extrahepatic cholangiocarcinoma or gallbladder cancer)
* Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST 1.1), as determined by the site investigator
* Participants with a history of hepatitis B or hepatitis C can be enrolled if they meet study criteria
* Is able to provide archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion
* Has a life expectancy of greater than 3 months
* Has adequate organ function

Exclusion Criteria

* Has had previous systemic therapy for advanced (metastatic) or unresectable (locally advanced) biliary tract cancer (intra-or extra hepatic cholangiocarcinoma or gallbladder cancer)
* Has ampullary cancer
* Has small cell cancer, neuroendocrine tumors, lymphoma, sarcoma, mixed tumor histology and/or mucinous cystic neoplasms
* Has received prior therapy with an anti-programmed cell death 1 (anti-PD-1), anti- programmed cell death ligand 1 or 2 (anti-PD-L1, anti-PD-L2) agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX-40, CD137)
* Has a known history of, or any evidence of, central nervous system (CNS) metastases and/or carcinomatous meningitis, as assessed by local site investigator
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2025-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (22):
- China (22):
  - Anhui Provincial Hospital ( Site 0140), Hefei, Anhui
  - Beijing Cancer Hospital ( Site 0138), Beijing, Beijing Municipality
  - Peking Union Medical College Hospital ( Site 0150), Beijing, Beijing Municipality
  - First Affiliated Hospital of The Third Military Medical University ( Site 0130), Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital ( Site 0154), Fuzhou, Fujian
  - 900 Hospital of the Joint ( Site 0137), Fuzhou, Fujian
  - Guangdong Provincial People s Hospital ( Site 0161), Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital ( Site 0133), Harbin, Heilongjiang
  - Hunan Provincial People Hospital ( Site 0142), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 0132), Changsha, Hunan
  - The Third Xiangya Hospital of Central South University ( Site 0157), Changsha, Hunan
  - The 81st Hospital of PLA ( Site 0128), Nanjing, Jiangsu
  - The First Hospital of Jilin University ( Site 0131), Changchun, Jilin
  - Zhongshan Hospital Fudan University ( Site 0129), Shanghai, Shanghai Municipality
  - Renji Hospital Shanghai Jiaotong University School of Medicine ( Site 0158), Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center ( Site 0160), Shanghai, Shanghai Municipality
  - Tangdu Hospital ( Site 0146), Xi’an, Shanxi
  - The First Affiliated Hospital of Xi an Jiaotong University ( Site 0145), Xi’an, Shanxi
  - West China Hospital of Sichuan University ( Site 0147), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital ( Site 0155), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital Zhejiang University ( Site 0136), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 0134), Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Yoo C, Ueno M, Klumpen HJ, Kelley RK, Vogel A, Furuse J, Ren Z, Yau T, Chan SL, Ozaka M, Oh SC, Gu S, Park JO, Valle JW, Edeline J, Kim JG, Kamble S, Norquist JM, Yu L, Malhotra U, Finn RS. Health-related quality of life in participants with advanced biliary tract cancer from the randomized phase III KEYNOTE-966 study. J Hepatol. 2025 Sep;83(3):692-700. doi: 10.1016/j.jhep.2025.03.019. Epub 2025 Mar 27. PMID 40154623
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://trialstransparency.merckclinicaltrials.com/Study.aspx?id=3475-966&kw=3475-966

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As of the data cut-off (DCO) (15-DEC-2022) for the final analysis (FA), a total of 158 participants were randomized to the Intent-to-Treat (ITT) population (75 in the pembrolizumab plus chemotherapy group and 83 in the placebo plus chemotherapy group)
Groups:
- Arm A (Pembrolizumab+Gemcitabine+Cisplatin): Pembrolizumab, 200 mg, every 3 weeks (Q3W), Day 1 of each 3-week cycle for up to 35 cycles PLUS Gemcitabine, 1000 mg/m^2, Q3W, Day 1 and Day 8 of each cycle until progressive disease or unacceptable toxicity PLUS Cisplatin, 25 mg/m^2, Q3W, Day 1 and Day 8 of each cycle for up to 8 cycles. Participants in Arm A who stopped study intervention after achieving stable-disease (SD) or better may have been eligible to receive additional pembrolizumab for up to 17 cycles if they experienced radiographic disease progression while off study intervention, according to the protocol-defined criteria. Gemcitabine may have been continued until progressive disease (PD) or unacceptable toxicity during second course at investigator's discretion.
Period: Overall Study
Arm/Group | Arm A (Pembrolizumab+Gemcitabine+Cisplatin) | Arm B (Placebo+Gemcitabine+Cisplatin)
Started | 75 | 83
Completed | 0 | 0
Not Completed | 75 | 83
Not completed — Death | 49 | 63
Not completed — Participant On-going | 26 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Pembrolizumab+Gemcitabine+Cisplatin) | Arm B (Placebo+Gemcitabine+Cisplatin) | Total
Number analyzed (Participants) | 75 | 83 | 158
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (8.3) | 58.6 (9.5) | 59.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 36 | 75
  Male | 36 | 47 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 75 | 83 | 158
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 75 | 83 | 158
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Geographic Region [Count of Participants; unit: Participants]
  Asian | 75 | 83 | 158
Disease Status [Count of Participants; unit: Participants]
  Locally Advance | 12 | 14 | 26
  Metastatic | 63 | 69 | 132
Site of Origin [Count of Participants; unit: Participants]
  Gallbladder | 19 | 12 | 31
  Intrahepatic | 45 | 60 | 105
  Extrahepatic | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from randomization to death due to any cause. Per protocol the final reported outcome for OS did not include any sensitivity or supportive analysis.
Time Frame: Up to approximately 29 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Pembrolizumab+Gemcitabine+Cisplatin) | Arm B (Placebo+Gemcitabine+Cisplatin)
Number analyzed (Participants) | 75 | 83
Months | 14.1 [10.4 to 17.7] | 9.9 [8.6 to 13.0]
Statistical Analysis 1: Comparison: Arm A (Pembrolizumab+Gemcitabine+Cisplatin) vs Arm B (Placebo+Gemcitabine+Cisplatin); Test type: Other; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.51 to 1.08] — HR=Arm A/Arm B

2. Secondary Outcome: Progression-free Survival (PFS) Per RECIST 1.1 as Assessed by BICR
Description: Progression-free survival was defined as the time from randomization to the first documented disease progression or death due to any cause, whichever occurred first.
Time Frame: Up to approximately 29 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Pembrolizumab+Gemcitabine+Cisplatin) | Arm B (Placebo+Gemcitabine+Cisplatin)
Number analyzed (Participants) | 75 | 83
Months | 5.6 [3.2 to 7.4] | 5.7 [4.4 to 6.9]
Statistical Analysis 1: Comparison: Arm A (Pembrolizumab+Gemcitabine+Cisplatin) vs Arm B (Placebo+Gemcitabine+Cisplatin); Test type: Other; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.58 to 1.19] — HR=Arm A/Arm B

3. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: ORR was defined as the percentage of participants who had a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: a ≥30% decrease in the sum of diameters [SOD] of target lesions) as assessed by BICR per RECIST 1.1, which was adjusted for this study to allow a maximum of 10 target lesions in total and 5 per organ.
Time Frame: Up to approximately 29 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Arm A (Pembrolizumab+Gemcitabine+Cisplatin) | Arm B (Placebo+Gemcitabine+Cisplatin)
Number analyzed (Participants) | 75 | 83
Percentage | 36.0 [25.2 to 47.9] | 28.9 [19.5 to 39.9]
Statistical Analysis 1: Comparison: Arm A (Pembrolizumab+Gemcitabine+Cisplatin) vs Arm B (Placebo+Gemcitabine+Cisplatin); Test type: Other; Difference in Percentages = 7.1, 95% CI 2-sided [-7.5 to 21.6] — Difference=Arm A minus Arm B

4. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR
Description: For participants who demonstrated a confirmed CR or PR, DOR was the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurred first.
Time Frame: Up to approximately 29 months
Population: All responders (participants that achieved complete or partial response)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Pembrolizumab+Gemcitabine+Cisplatin) | Arm B (Placebo+Gemcitabine+Cisplatin)
Number analyzed (Participants) | 27 | 24
Months | 10.2 [5.4 to NA] — Upper limit not reached | 5.7 [4.2 to 14.0]

5. Secondary Outcome: Number of Participants Who Experience One or More Adverse Events (AE)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it was considered related to the medical treatment or procedure, that occurred during the course of the study.
Time Frame: Up to approximately 29 months
Population: All Participants as Treated (APaT) population, which consisted of all randomized participants who received at least 1 dose of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Pembrolizumab+Gemcitabine+Cisplatin) | Arm B (Placebo+Gemcitabine+Cisplatin)
Number analyzed (Participants) | 74 | 82
Participants | 73 | 82

6. Secondary Outcome: Number of Participants Who Discontinued Study Intervention Due to an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it was considered related to the medical treatment or procedure, that occurred during the course of the study.
Time Frame: Up to approximately 29 months
Population: APaT population, which consisted of all randomized participants who received at least 1 dose of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Pembrolizumab+Gemcitabine+Cisplatin) | Arm B (Placebo+Gemcitabine+Cisplatin)
Number analyzed (Participants) | 74 | 82
Participants | 18 | 14

ADVERSE EVENTS:
Time Frame: Up to approximately 29 months
Description: All-Cause Mortality included all allocated participants. Serious and Other AEs were reported according to treatment course for all participants who received ≥1 dose of study treatment. As of DCO (15-DEC-2022) for the FA, none of the participants received the optional 2nd course of treatment.
Groups:
- Pembrolizumab + Chemotherapy First Course: Pembrolizumab, 200 mg, every 3 weeks (Q3W), Day 1 of each 3-week cycle for up to 35 cycles PLUS Gemcitabine, 1000 mg/m^2, Q3W, Day 1 and Day 8 of each cycle until progressive disease or unacceptable toxicity PLUS Cisplatin, 25 mg/m^2, Q3W, Day 1 and Day 8 of each cycle for up to 8 cycles.
- Placebo + Chemotherapy First Course: Placebo to Pembrolizumab, 200 mg, every 3 weeks (Q3W), Day 1 of each 3-week cycle for up to 35 cycles PLUS Gemcitabine, 1000 mg/m^2, Q3W, Day 1 and Day 8 of each cycle until progressive disease or unacceptable toxicity PLUS Cisplatin, 25 mg/m^2, Q3W, Day 1 and Day 8 of each cycle for up to 8 cycles.
Arm/Group | Pembrolizumab + Chemotherapy First Course | Placebo + Chemotherapy First Course
All-Cause Mortality (participants affected / at risk) | 49/75 | 63/83
Serious Adverse Events (participants affected / at risk) | 28/74 | 29/82
Other Adverse Events (participants affected / at risk) | 73/74 | 82/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Chemotherapy First Course (N=74) | Placebo + Chemotherapy First Course (N=82)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (2)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 5 (5)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 4 (6) | 4 (4)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Myocardial necrosis marker increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (6) | 2 (2)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 9 (9) | 7 (11)
White blood cell count decreased (Investigations) | 3 (3) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Chemotherapy First Course (N=74) | Placebo + Chemotherapy First Course (N=82)
Anaemia (Blood and lymphatic system disorders) | 59 (101) | 65 (100)
Hyperthyroidism (Endocrine disorders) | 4 (4) | 2 (2)
Hypothyroidism (Endocrine disorders) | 11 (13) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 7 (10) | 8 (10)
Abdominal pain (Gastrointestinal disorders) | 5 (10) | 6 (7)
Abdominal pain upper (Gastrointestinal disorders) | 6 (9) | 11 (22)
Ascites (Gastrointestinal disorders) | 0 (0) | 7 (7)
Constipation (Gastrointestinal disorders) | 15 (26) | 20 (30)
Diarrhoea (Gastrointestinal disorders) | 12 (16) | 5 (7)
Nausea (Gastrointestinal disorders) | 38 (97) | 35 (88)
Vomiting (Gastrointestinal disorders) | 31 (82) | 37 (88)
Asthenia (General disorders) | 14 (40) | 11 (25)
Chest discomfort (General disorders) | 5 (6) | 5 (6)
Fatigue (General disorders) | 5 (5) | 7 (7)
Malaise (General disorders) | 12 (21) | 11 (20)
Oedema peripheral (General disorders) | 5 (5) | 5 (7)
Pyrexia (General disorders) | 11 (16) | 10 (17)
Hepatic function abnormal (Hepatobiliary disorders) | 5 (16) | 6 (11)
Hepatic pain (Hepatobiliary disorders) | 4 (5) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 5 (6)
Alanine aminotransferase increased (Investigations) | 16 (27) | 28 (45)
Aspartate aminotransferase increased (Investigations) | 19 (36) | 30 (57)
Blood alkaline phosphatase increased (Investigations) | 11 (11) | 8 (10)
Blood bilirubin increased (Investigations) | 9 (10) | 15 (24)
Blood creatinine increased (Investigations) | 3 (10) | 9 (20)
Blood lactate dehydrogenase increased (Investigations) | 5 (9) | 6 (21)
Gamma-glutamyltransferase increased (Investigations) | 8 (13) | 12 (18)
Lymphocyte count decreased (Investigations) | 13 (35) | 13 (26)
Neutrophil count decreased (Investigations) | 55 (328) | 58 (316)
Neutrophil count increased (Investigations) | 4 (8) | 1 (2)
Platelet count decreased (Investigations) | 47 (211) | 46 (152)
Total bile acids increased (Investigations) | 4 (5) | 6 (10)
Weight decreased (Investigations) | 10 (10) | 14 (19)
Weight increased (Investigations) | 4 (4) | 6 (6)
White blood cell count decreased (Investigations) | 58 (376) | 62 (323)
Decreased appetite (Metabolism and nutrition disorders) | 20 (47) | 28 (56)
Electrolyte imbalance (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (9) | 8 (11)
Hyperuricaemia (Metabolism and nutrition disorders) | 9 (41) | 11 (21)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (13) | 16 (27)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (3) | 6 (8)
Hypochloraemia (Metabolism and nutrition disorders) | 2 (5) | 10 (16)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (15) | 13 (18)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (13) | 12 (28)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (17) | 15 (21)
Hypoproteinaemia (Metabolism and nutrition disorders) | 3 (3) | 6 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (6)
Dizziness (Nervous system disorders) | 3 (3) | 8 (9)
Headache (Nervous system disorders) | 5 (7) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (4) | 5 (5)
Renal impairment (Renal and urinary disorders) | 4 (9) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (12) | 11 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 15 (19) | 8 (15)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 5 (10)
Thrombosis (Vascular disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agreed to submit all manuscripts or abstracts to the Sponsor before submission. This allowed the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT04924062/Prot_SAP_001.pdf